CLINICAL TRIAL: NCT07198464
Title: A Prospective, Multicenter Clinical Study of Relmacabtagene Autoleucel Combined With Autologous Hematopoietic Stem Cell Transplantation, Orelabrutinib, and Sintilimab for Primary Central Nervous System Lymphoma
Brief Title: Relmacabtagene Autoleucel Combined With Autologous Hematopoietic Stem Cell Transplantation, Orelabrutinib, and Sintilimab for Primary Central Nervous System Lymphoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Mingzhi Zhang, Department Director, Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-ZD-003-ATT02
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL)
MeSH Terms: interventions — relmacabtagene autoleucel; Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- relmacabtagene autoleucel and transplantation (Experimental): relmacabtagene autoleucel combined with autologous hematopoietic stem cell transplantation, with orelabrutinib, and sintilimab as maintenance therapy
  Interventions: Drug: Relmacabtagene autoleucel and transplantation

INTERVENTIONS:
Drug: Relmacabtagene autoleucel and transplantation — This study enrolled patients with primary central nervous system lymphoma, from whom mononuclear cells and hematopoietic stem cells were collected. Participants receive infusions of hematopoietic stem cells and CAR-T cells, followed by maintenance therapy with orelabrutinib and sintilimab starting on day 15 post-transplantation, for a median duration of up to 6 months and 1 year, respectively.

SUMMARY:
To evaluate the efficacy and safety of relmacabtagene autoleucel combined with autologous hematopoietic stem cell transplantation, orelabrutinib, and sintilimab as first-line or relapsed/refractory treatment for primary central nervous system diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1.18-60 years 2.ECOG performance status 0-2 3.No prior treatment with CAR-T cell therapy or autologous stem cell transplantation (ASCT) 4.Expected survival ≥ 3 months 5.No history of malignancy (except for in situ carcinoma or other indolent malignancies), or inactive malignancy with treatment completed >1 year ago 6.Histopathologically confirmed PCNSL (lymphoma confined to the brain without systemic involvement, with histopathological type being diffuse large B-cell lymphoma, or systemic lymphoma with central nervous system involvement and histopathological type being diffuse large B-cell lymphoma) 7.Refractory disease is defined as failure to achieve complete remission after first-line therapy (excluding intolerance to first-line therapy), including: Progressive disease (PD) as best response to first-line therapy, or Stable disease (SD) as best response after at least 4 cycles of first-line therapy (e.g., 4 cycles of R-CHOP), or Residual disease after at least 6 cycles of first-line therapy, or relapse within 12 months after completing first-line therapy 8.Relapsed disease is defined as recurrence after achieving complete remission following first-line therapy, occurring within 12 months after treatment completion 9.Positive CD19 expression by immunohistochemistry 10.No contraindications for CAR-T cell therapy or ASCT 11.No concurrent use of other anti-tumor therapies during this treatment; bisphosphonates for bone metastases and symptomatic supportive treatments are allowed 12.Able to understand the study and provide signed Informed Consent Form

Exclusion Criteria:

1. Pregnant or lactating women
2. Any uncontrolled medical condition (including active infection, uncontrolled diabetes, severe cardiac, hepatic or renal insufficiency, interstitial pneumonia, etc.)
3. Use of systemic corticosteroids within 7 days before CD19 CAR-T cell infusion (except ≤ 5 mg/day dexamethasone or equivalent doses of other corticosteroids)
4. Prior exposure to ≥ 2 of the following agents with documented resistance: orelabrutinib, fotemustine, carmustine, thiotepa, or PD-1/PD-L1 inhibitors
5. History of autoimmune disease
6. Presence of cachexia or any other contraindication to chemotherapy
7. Active, uncontrolled infection
8. History of poorly controlled psychiatric disorder
9. Any condition that, in the opinion of the investigator, would preclude safe participation in this trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-07 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival(PFS) | Up to 60 months
  PFS is defined as the time from CAR-T infusion to the first occurrence of either disease progression or death from any cause, whichever comes first, regardless of whether study treatment has been discontinued prior to the PFS event.
overall response rate(ORR) | Up to 3 months

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 60 months